CLINICAL TRIAL: NCT01970553
Title: Phase I Multicenter, Open-label, Clinical and Pharmacokinetic Study of PM01183 in Combination With Gemcitabine in Non-heavily Pretreated Patients With Selected Advanced Solid Tumors
Brief Title: Escalating Doses of PM01183 in Combination With Gemcitabine in Patients With Specific Unresectable Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM1183-A-004-10
Record Dates: First submitted 2013-10-22; First posted 2013-10-28 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2013-10

CONDITIONS: Specific Advanced Solid Tumors
Keywords: lurbinectedin; PM01183; tumors; cancer; Pharma Mar
MeSH Terms: conditions — Neoplasms | interventions — PM 01183; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lurbinectedin (PM01183) / gemcitabine (Experimental): Patients will consecutively receive the following on Days 1 and 8 q3wk (three weeks = one treatment cycle):
  - Gemcitabine: intravenous infusion of 800 mg/m2/day over 30 minutes,
  immediately followed by:
  - PM01183: intravenous infusion over one hour at a starting dose of 2.5 mg/day, flat dose (FD), both on Days 1 and 8 every 3 weeks
  Interventions: Drug: lurbinectedin (PM01183); Drug: Gemcitabine

INTERVENTIONS:
Drug: lurbinectedin (PM01183) — lurbinectedin (PM01183) is presented as powder for concentrate for solution for infusion with two strengths, 1-mg and 4-mg vials
Drug: Gemcitabine — 1000 mg vial, powder for injectable solution

SUMMARY:
Phase I multicenter, open-label, clinical and pharmacokinetic study of PM01183 in combination with gemcitabine in non-heavily pretreated patients with selected advanced solid tumors to determine the maximum tolerated dose (MTD) and the recommended dose (RD) of PM01183 in combination with gemcitabine, to characterize the safety profile and feasibility of this combination in patients with selected advanced solid tumors, to characterize the pharmacokinetics (PK), to obtain preliminary information on the clinical antitumor activity in non-heavily pretreated selected solid tumor patients and to evaluate the pharmacogenomics (PGx) in tumor samples of patients exposed, in order to assess potential markers of response and/or resistance.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily written informed consent
* Age: between 18 and 75 years (both inclusive)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 1
* Life expectancy ≥ 3 months
* Patients with a histologically/cytologically confirmed diagnosis of advanced disease of any of the following tumors:

  1. Breast cancer
  2. Epithelial ovarian cancer (including primary peritoneal disease and/or fallopian tube carcinomas and/or endometrial adenocarcinomas)
  3. Stromal uterine sarcomas
  4. Non-small cell lung cancer (NSCLC)
  5. Platinum-refractory or relapsed germ cell tumors
  6. Adenocarcinoma of the exocrine pancreas
  7. Biliary tract adenocarcinoma
  8. Adenocarcinoma or carcinoma of unknown primary site
  9. Advanced or unresectable mesothelioma
* At least three weeks since the last anticancer therapy,including radiation therapy (RT)
* Adequate bone marrow, renal, hepatic, and metabolic function
* Left ventricular ejection fraction (LVEF) by echocardiography (ECHO) or multiple-gated acquisition (MUGA) within normal range (according to institutional standards).
* Women of childbearing potential must have a negative serum pregnancy test before study entry. Both women and men must agree to use a medically acceptable method of contraception throughout the treatment period and for six weeks after discontinuation of treatment.

Exclusion Criteria:

* Concomitant diseases/conditions:

  * History or presence of unstable angina, myocardial infarction, congestive heart failure, or clinically significant valvular heart disease within last year.
  * Symptomatic or any uncontrolled arrhythmia
  * Ongoing chronic alcohol consumption, or cirrhosis
  * Active uncontrolled infection.
  * Known human immunodeficiency virus (HIV) infection.
  * Any other major illness that, in the Investigator's judgment
* Brain metastases or leptomeningeal disease involvement
* Men or women of childbearing potential who are not using an effective method of contraception
* Patients who have had radiation therapy in more than 35% of the bone marrow
* History of previous bone marrow and/or stem cell transplantation
* Prior treatment with gemcitabine-containing therapy for advanced disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2011-05; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Recommended Dose (RD) | 19 months
  The RD will be the highest dose level explored at which less than one third of evaluable patients experience a DLT during Cycle 1.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) characterisation | 19 months
  The dose-exposure relationships for maximum plasma concentration (Cmax) and area under the curve (AUC) will be evaluated.
Preliminary antitumor efficacy | 29 months
  To obtain preliminary information on the clinical antitumor activity of this combination in non-heavily pretreated selected solid tumor patients
Pharmacogenomics (PGx) | 29 months
  to identify molecular markers whose expression may be associated with the clinical outcome of patients. These molecular markers might allow the identification of those patients who will benefit from PM01183 and gemcitabine treatment, thus improving the health care by an individualized medicine.

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Szyldergemajn, MD, Study Chair — Pharma Mar
Locations (3):
- Spain (2):
  - Hospital Universitario Madrid Sanchinarro, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
- University College of London Hospital, London, United Kingdom